CLINICAL TRIAL: NCT07056387
Title: The Effects of a Nurse-led Community-based Sailing Programme on Resilience of School-aged Children With Autism: A Randomised Controlled Trial
Brief Title: The Effects of a Nurse-led Community-based Sailing Programme on Resilience of School-aged Children With Autism: An RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Sailability Hong Kong (Unknown)
Responsible Party: Principal Investigator, Myrian Sze Nga Fan, PhD Candidate, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC 2025.237-T
Record Dates: First submitted 2025-06-29; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Autism Spectrum Disorder; Resilience
Keywords: Sailing; Nature-based interventions; School-aged children
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The intervention is guided by the Synergy Model of Resilience, integrating Kolb's theory of experiential learning.
Who Masked: Outcomes Assessor
Masking Description: The study employs single masking, where only the outcome assessor is blinded. Due to the nature of the interventions, masking the participants and intervention providers is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Eligible participants will participate in the nurse-led CBS programme, utilising dinghies with a universal design known for their exceptional stability to prioritize safety. The concrete experience will be introduced through sailing activities. The instructor-to-participant ratio will be 1:6 with a safety boat present.
  Interventions: Other: A nurse-led community-based sailing programme
- Attention controlled Group (Active Comparator): The attention control group participates in crafting activities (e.g., making handicrafts or painting) to engage participants in an active process, allowing for a comparison of the intervention's effects (sailing programme) against an alternative active activity.
  Interventions: Other: Crafting activities

INTERVENTIONS:
Other: A nurse-led community-based sailing programme — A nurse-led community-based sailing programme is validated by an expert panel including professionals from various fields, such as a registered nurse, academia, and qualified sailing instructors, delivered in a group of 6 participants, incorporating experiential learning, with the aid of materials including dinghies with Universal design, safety boats, buoys, buoyancy aids, supplementing with a waterproof sailing booklet. The intervention is developed and facilitated by a registered nurse (principal investigator).
  Arms: Intervention group
Other: Crafting activities — Participants in the attention control group will participate in crafting activities. Activities match the time and attention dedicated by the intervention group. Activities are designed to have no impact on resilience.
  Arms: Attention controlled Group

SUMMARY:
The goal of this randomised controlled trial is to evaluate the effect of a nurse-led community-based sailing programme on resilience of school-aged children with autism in inclusive education.

Does intervention improve the resilience of participants? Does intervention improve the quality of life, self-esteem, depressive symptoms, and social functioning outcomes of participants?

Researchers will compare the effect of intervention (community-based sailing programme) to the attention control group (Crafting activities) at baseline, post-intervention, and at 3-month and 9-month follow-ups.

Participants will:

Participants in the intervention group will participate in a nurse-led community-based sailing programme over six days, with each day consisting of 4 sessions, each lasting an hour, for a total of 24 hours.

Participants in the attention control group will engage in crafting activities with minimal difficulty, focusing on maintaining attention without any emotional or reflective discussions.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental condition that typically emerges in early childhood, characterized by persistent deficits in social communication and interaction, with the presence of restricted, repetitive patterns of behaviour, interests, or activities. This study seeks to address the outcome gap in the literature, the resilience of children with ASD, and contribute to their holistic health through integrating nature and the community.

The study hypothesizes that, compared to the attention control group, school-aged children with ASD in inclusive education who participate in the intervention group will exhibit: (1) increased levels of resilience, (2) improved quality of life (QoL), (3) reduced depressive symptoms, (4) enhanced self-esteem, and (5) improved social functioning, both immediately post-intervention and at 3-month and 9-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 7 and 12,
* Have a confirmed diagnosis of ASD,
* Be enrolled in an inclusive education school,
* Possess the ability to complete the questionnaire in Chinese,
* Be able to communicate in Chinese.

Exclusion Criteria:

* With sailing experience,
* With a history of severe motion sickness symptoms.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Resilience | Pre-intervention, Post-intervention (within 1 week immediately after intervention), and at 3-month and 9-month follow-ups.
  Resilience will be measured using the 14-item Resilience Scale (RS-14), which assesses personal competence, self-acceptance, and life acceptance. Each item is rated on a 7-point Likert scale (1 = "strongly disagree" to 7 = "strongly agree"), with total scores ranging from 14 to 98. Higher scores indicate greater resilience. The validated Chinese version of the RS-14, with a Cronbach's alpha of 0.86, has demonstrated good internal consistency for assessing resilience in young adolescents in Hong Kong.

SECONDARY OUTCOMES:
Depressive symptoms | Pre-intervention, Post-intervention (within 1 week immediately after intervention), and at 3-month and 9-month follow-ups.
  Depressive symptoms will be assessed using the Chinese version of the Center for Epidemiologic Studies Depression Scale for Children (CES-DC). The scale includes 20 items across emotional, cognitive, and behavioral domains of depression. Participants rate the frequency of symptoms over the past week on a 4-point Likert scale (0 = not at all, 1 = a little, 2 = some, 3 = a lot). Total scores range from 0 to 60, with higher scores indicating more severe depressive symptoms. A score of 16 or higher suggests the presence of depressive symptoms. The Chinese version of the CES-DC, validated for use in children in Hong Kong, demonstrates strong internal consistency (Cronbach's alpha > 0.8).
Self-esteem | Pre-intervention, Post-intervention (within 1 week immediately after intervention), and at 3-month and 9-month follow-ups.
  Self-esteem will be measured using Rosenberg's Self-Esteem Scale (RSES), a validated tool for assessing global self-worth. The scale comprises 10 items, rated on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree). Total scores range from 10 to 40, with higher scores reflecting higher levels of self-esteem. The Chinese version of the RSES has been validated in Hong Kong, showing good internal consistency (Cronbach's alpha = 0.78).
Quality of life (QoL) | Pre-intervention, Post-intervention (within 1 week immediately after intervention), and at 3-month and 9-month follow-ups.
  QoL will be assessed using the Pediatric Quality-of-Life Inventory 4.0 Generic Core Scale (PedsQL™). This 23-item questionnaire evaluates physical functioning (8 items), emotional functioning (5 items), social functioning (5 items), and school functioning (5 items). Participants rate the extent of problems experienced in the past month on a 5-point Likert scale (0 = never to 4 = almost always). Scores are reverse-coded and linearly transformed to a 0-100 scale, with higher scores indicating better QoL. The Chinese version of the PedsQL™, validated in Hong Kong, demonstrates excellent internal consistency (Cronbach's alpha = 0.90).
Social functioning outcomes | Pre-intervention, Post-intervention (within 1 week immediately after intervention), and at 3-month and 9-month follow-ups.
  Social functioning will be evaluated using the 2nd edition of the Social Responsiveness Scale (SRS-2), a 65-item questionnaire assessing ASD-related symptoms. Participants' parents rate each item on a 4-point Likert scale (0 = never true to 3 = almost always true). The SRS-2 includes five subscales: social awareness, social cognition, social communication, social motivation, and autistic mannerisms, as well as a total score. Higher scores indicate greater impairment in social functioning. The Chinese version of the SRS-2 has been validated in China, showing strong internal consistency (Cronbach's alpha = 0.90).

CONTACTS AND LOCATIONS:
Overall Officials: Myrian Sze Nga Fan, MSc, Principal Investigator — Chinese University of Hong Kong; William Ho Cheung Li, PhD, Study Director — Chinese University of Hong Kong; Laurie Long Kwan Ho, PhD, Study Director — Chinese University of Hong Kong; Sek Ying Chair, PhD, Study Chair — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No
The research team does not have plans to proactively or automatically make the individual participant data (IPD) from this study available to other researchers. However, the IPD may be shared upon request, provided that the requesting party has a valid scientific or medical rationale and obtains the necessary approval from the research team.
  Any requests for access to the study's IPD will be reviewed on a case-by-case basis by the research team. Factors that will be considered in evaluating such requests include:
  * Scientific merit and validity of the proposed use of the data
  * Qualifications and track record of the requesting researcher or research team
  * Alignment with the original study objectives and participants' consent